CLINICAL TRIAL: NCT07045116
Title: Effectiveness of Electronic Anesthesia Delivery Syringe Versus Conventional Syringe on Pain and Anxiety Perception During Local Anesthetic Injection in Children Randomized Clinical Trial
Brief Title: Electronic vs. Conventional Syringes: Impact on Pediatric Pain and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Randa Omer Ahmed Bashir (Other)
Responsible Party: Sponsor-Investigator, Randa Omer Ahmed Bashir, Master's degree candidate at Pediatric department, Ain Shams University, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: FDASU-Rec IM012410
Record Dates: First submitted 2025-05-28; First posted 2025-07-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-12

CONDITIONS: Dental Anxiety; Pain Management
Keywords: dental anxiety; salivary amylase; dental syringes; electronic anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: In our dental study, the investigator will utilize a computerized system called "Sealed Envelope" to implement a random assignment of the treatment options of the participants' teeth. This randomization process is crucial to ensure that each participant receives either conventional or electronic anesthesia during their first dental treatment. While, during their second dental treatment the alternative method of anesthesia will be used.
  The trial is specifically constructed such that for each participant, electronic anesthetic will be applied to teeth on the right side, whereas conventional anesthesia will be used on the left side.
  To uphold the principles' allocation concealment, which is essential for maintaining the study's integrity. It will be kept with a third party, who will not be involved in the data collection. The allocation assignment of the participants will be requested each time a new participant is recruited in the trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary right primary molar (Active Comparator): Maxillary right primary molar will receive electronic anesthesia
  Interventions: Device: Electronic anesthesia
- Maxillary left primary molar (Active Comparator): Maxillary left primary molar will receive conventional anesthesia
  Interventions: Device: Conventional anesthesia

INTERVENTIONS:
Device: Electronic anesthesia — The child will receive electronic anesthesia to the right side of the upper jaw; the pain and anxiety level will be assessed.
  Other Names: pen injector
  Arms: Maxillary right primary molar
Device: Conventional anesthesia — The child will receive conventional anesthesia to the maxillary left side
  Other Names: Conventional syringe
  Arms: Maxillary left primary molar

SUMMARY:
Study Overview Purpose: To compare pain and anxiety levels in children aged 6-8 during local anesthesia administration using electronic vs. conventional syringes.

Design: Split-mouth randomized controlled trial (RCT) involving 40 children receiving both types of anesthesia during pulp therapy of bilateral maxillary primary molars.

Objectives Primary Outcome: Pain level measured via Visual Analogue Scale (VAS).

Secondary Outcomes:

Physiological markers: heart rate and oxygen saturation via pulse oximetry.

Salivary amylase levels (anxiety biomarker) assessed using ELISA.

Methodology Children are randomly assigned to receive electronic anesthesia on one side and conventional on the other in two separate visits.

Saliva samples are collected before and after each injection.

Double-blind setup: children blinded using sunglasses; statistician also blinded.

Same operator administers all injections for consistency.

Ethical Considerations Written informed consent and assent obtained.

Risks (e.g., systemic toxicity, allergic reactions) minimized via dosage limits and patient monitoring.

Privacy and data security measures in place.

Statistical Analysis Data analyzed using SPSS; significance set at p ≤ 0.05.

Sample size calculated for adequate power (n = 33 minimum; 40 enrolled).

Funding Self-funded.

Clinical Relevance Electronic anesthesia may offer a less painful and anxiety-inducing alternative for pediatric dental patients, potentially improving children's long-term attitude toward dental care.

DETAILED DESCRIPTION:
1. Title and Context Title: Effectiveness of Electronic Anesthesia Delivery Syringe Versus Conventional Syringe on Pain and Anxiety Perception During Local Anesthetic Injection in Children.

   Submitted by: Randa Omer Ahmed Bashir, for partial fulfillment of a master's degree in Pediatric Dentistry at Ain Shams University.

   Supervisors: Assoc. Prof. Dr. Reham Khaled Elghazawy and Dr. Nour Abdelmonem Wahba.
2. Abstract Problem Statement: Local anesthesia causes pain and anxiety, especially in children.

   Objective: To compare electronic vs. conventional anesthesia during pulp therapy in 6-8-year-old children.

   Design: Split-mouth RCT involving 40 children.

   Outcomes:

   Primary: Pain measured by Visual Analogue Scale (VAS).

   Secondary: Heart rate, oxygen saturation, and salivary amylase (stress biomarker) using ELISA.
3. Background Local anesthesia is a primary source of fear in children due to needle insertion, pressure, and speed of delivery.

   Minimizing pain and anxiety is critical for long-term positive dental attitudes.

   Electronic anesthesia devices may reduce these discomforts through:

   Controlled delivery rate.

   Reduced injection pressure.

   Numbing tissue ahead of the needle.
4. Research Question (PICOTS Framework) Population: 40 children (6-8 years old).

   Intervention: Electronic anesthesia.

   Comparator: Conventional anesthesia.

   Outcome: Pain (VAS), heart rate, oxygen saturation, salivary amylase.

   Time: Two visits.

   Setting: Ain Shams University Pediatric Dentistry outpatient clinic (Jan 2024-Jan 2025).
5. Aim and Objectives Aim: To assess pain and anxiety levels during local anesthesia using electronic vs. conventional syringes.

   Primary Outcome:

   Pain via VAS before and after anesthesia.

   Secondary Outcomes:

   Heart rate and oxygen saturation using pulse oximetry.

   Salivary amylase levels via ELISA test.
6. Hypothesis Null Hypothesis (H0): No difference between electronic and conventional anesthesia in reducing pain and anxiety.
7. Ethical Considerations Risks: Pain, discomfort, self-injury post-procedure, potential allergic reactions.

   Risk Minimization:

   Proper selection and dosage of anesthetic agents.

   Use of topical anesthetic pre-injection.

   Postoperative instructions to avoid tissue trauma.

   Privacy & Confidentiality: Anonymized data using patient codes.

   Informed Consent: Written consent and assent obtained.

   Adverse Events: Monitored and reported with defined procedures.

   Sample Disposal: Discarded as biohazardous waste after study completion.
8. Study Design Type: Randomized Controlled Trial (RCT).

   Design: Split-mouth, double-blinded.

   Blinding:

   Patients blinded with sunglasses.

   Statistician and assessors blinded to allocation.

   Randomization Tool: Sealed Envelope computer-generated randomization.

   Allocation Concealment: Handled by a third party.
9. Materials and Methods Study Population

   Inclusion Criteria:

   6-8 years old.

   Medically free (ASA I).

   First dental visit.

   At least one vital deep carious molar on each side of maxilla.

   Exclusion Criteria:

   Allergy to local anesthetic.

   Use of corticosteroids or drugs affecting saliva.

   Declined consent.

   Sample Size:

   Required Sample: 33 children (based on power analysis).

   Final Enrolled: 40 children.

   Intervention Procedures:

   Visit 1:

   One side receives either conventional or electronic anesthesia according to randomization.

   (Fact: the right side always received electronic anesthesia, while the left side received conventional anesthesia).

   Visit 2:

   Opposite side receives the other type of anesthesia.

   Procedure:

   Topical anesthetic applied 1-2 minutes.

   Injection using 4% articaine with 1:100,000 adrenaline.

   VAS recorded post-injection.

   Heart rate and oxygen saturation measured pre- and post-injection using pulse oximeter.

   Saliva samples collected:

   Pre-injection (baseline).

   Post-injection (after each type).

   Saliva stored frozen and tested with ELISA.
10. Bias Minimization Strategies Selection Bias: Controlled through randomization and allocation concealment.

    Performance Bias: Double-blind design.

    Detection Bias: Blinded outcome assessors.

    Attrition Bias: Risk due to single follow-up, acknowledged in design.

    Reporting Bias: All outcomes will be reported.
11. Statistical Analysis Software: IBM® SPSS® Statistics Version 26.

    Tests:

    Categorical data: Chi-square test.

    Numerical data:

    Normal distribution: Mean ± SD, Paired t-test.

    Non-normal distribution: Median and range, Wilcoxon signed-rank test.

    Significance Level: p ≤ 0.05.
12. Funding Source: Self-funded.
13. Clinical Relevance Electronic anesthesia offers less pain, better anxiety control, and may become a preferred technique in pediatric dentistry, especially for first-time dental patients.

ELIGIBILITY:
Inclusion Criteria:

* 6-8-year-old children.
* Medically free (ASA class I).
* Children attending their first dental visit.
* The patient should have at least one vital primary molar with deep carious lesion on each side.

Exclusion Criteria:

* Patient has any allergy to local anesthesia.
* Patients take any medications that affect the salivary flow.
* Patient taken corticosteroid.
* Children whose parents or legal guardians refuse to sign the informed consent.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Pain Perception | Timing: Immediately after the administration of local anesthesia (both electronic and conventional)
  Tool: Visual Analogue Scale (VAS)
  Scale: 0 (no pain) to 10 (worst possible pain)
  Purpose: To quantitatively assess the child's subjective pain level post-injection.

SECONDARY OUTCOMES:
Heart Rate (HR) | Immediately before and after the administration of local anesthesia (both electronic and conventional)
  Using Finger-type Pulse Oximeter
Oxygen Saturation | Immediately before and after both the Electronic and Conventional anesthesia
  Using Finger-type Pulse Oximeter
Salivary amylase level | Before any injection (baseline) - After conventional anesthesia (The saliva samples must be collected up to 30 minutes after the injection) - After electronic anesthesia (The saliva samples must be collected up to 30 minutes after the injection)
  Using ELIZA kit (Enzyme-Linked Immunosorbent Assay)

CONTACTS AND LOCATIONS:
Overall Officials: Reham Khaled Elghazawy, Associate professor, Study Director — Faculty of Dentistry, Ain Shams university; Nour Wahba, Lecturer/ Pedodontist, Study Director — Faculty of Dentistry, Ain Shams university
Locations (1):
- Faculty of Dentistry, Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The Ethical committee refuse to share the patient information because of confidentiality